CLINICAL TRIAL: NCT02740725
Title: The Role of Interactive Binocular Treatment System in Amblyopia Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamideh Sabbaghi, Shahid Beheshti Medical University, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sbmu.rec.1393.591
Record Dates: First submitted 2016-04-06; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Amblyopia
Keywords: Amblyopia; Interaction Binocular Treatment (I-BiTTM); Patch Therapy
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Recommendation of Patching (Active Comparator): Patients will receive two hours of patching in the case of one line difference of best corrected visual acuity(BCVA) between two eyes during one month.
  Interventions: Other: Patching Therapy
- Recommendation of Patching and interactive binocular treatment (Active Comparator): Patients will receive interactive binocular treatment addition to patch therapy in the least of 4 to 5 days of a week within 20-30 minutes in each day during one month.
  Interventions: Other: Patching Therapy; Device: Interactive Binocular Treatment System

INTERVENTIONS:
Other: Patching Therapy — Occlusion of a dominant eye with better best corrected visual acuity
Device: Interactive Binocular Treatment System — Dissociation of two eyes with more foveal stimulation to the amblyopic eye
  Arms: Recommendation of Patching and interactive binocular treatment

SUMMARY:
Purpose: of determining the role of Interactive Binocular Treatment (I-BiTTM) as a complementary method of patching in amblyopia therapy.

Materials and Methods: In this randomized clinical trial study, 50 unilateral amblyopic children (25 male/25 female) less than 10 years with either best corrected visual acuity (BCVA) ≤0.3 LogMAR (Logarithm minimum angle of resolution) in amblyopic eye or difference of VA≥2 lines between two eyes will be included. Patients will be classified in the case and control groups (25 in each), randomly. Patching will be recommended in both, cases will also received I-BiTTM. The child will be asked to play I-BiTTM games through glasses with conjugate colored filters. Patching was continued for one month more in both groups. VA and stereoacuity were measured at baseline, one month at the end of I-BiTTM treatment and one month after I-BiTTM treatment.

DETAILED DESCRIPTION:
In this clinical trial study, our case group will receive I-BiTTM in the format of three playing games which have been designed suitable to the age of our cases. The mechanism of I-BiTTM has been designed in three playing games with inducing more foveal stimulation for the amblyopic eye through presentation of movable targets with more detailed. In addition, unmovable targets will presented to the non-amblyopic eyes. Playing games were continued 30 minutes in each session for 5 days in each week within one month.

ELIGIBILITY:
Inclusion Criteria:

* BCVA <= 0.3 LogMAR

Exclusion Criteria:

* Organic Amblyopia
* Age less than 4 years
* Nystagmus

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity, Stereopsis | 30 days
  Two arms were under patching and Interactive Binocular Treatment (IBIT)

CONTACTS AND LOCATIONS:
Overall Officials: Zhale Rajavi, Professor, Study Director — Ophthalmic Research Center, Shahid Beheshti University of Medical Sciences, Tehran, Iran.
Locations (1):
- Islamic Republic of Iran, Tehran, Iran

REFERENCES:
- [Derived] Rajavi Z, Sabbaghi H, Amini Sharifi E, Behradfar N, Yaseri M. The role of Interactive Binocular Treatment system in amblyopia therapy. J Curr Ophthalmol. 2016 Aug 9;28(4):217-222. doi: 10.1016/j.joco.2016.07.005. eCollection 2016 Dec. PMID 27830207